CLINICAL TRIAL: NCT01193010
Title: Computer-Assisted Versus Non-Computer Assisted Preoperative Planning of Corrective Osteotomy for Extra-Articular Distal Radius Malunions: A Multi-Center Randomized Controlled Trial
Brief Title: Computer Assisted Planing of Corrective Osteotomy for Distal Radius Malunion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AO foundation (Unknown)
Responsible Party: Principal Investigator, Jesse B. Jupiter, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010P000444
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Extraarticular Distal Radius Malunion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Surgery without computer-assisted planning.
  Interventions: Procedure: distal radius osteotomy
- Computer-Assisted Surgical Planning (Experimental)
  Interventions: Procedure: Computer-Assisted Surgical Planning

INTERVENTIONS:
Procedure: Computer-Assisted Surgical Planning — Using a CT reconstructing of affected distal radius and the normal contralateral limb, surgical guides for the osteotomy will be created to assist with surgical planning.
  Arms: Computer-Assisted Surgical Planning
Procedure: distal radius osteotomy — In this control group, the planning and surgical execution of the distal radius osteotomy will be performed as usual, without computer-assisted planning of the osteotomy.
  Arms: Control

SUMMARY:
This study is designed as a multi-center randomized controlled trial, comparing two groups of patients with symptomatic extra-articular malunited distal radius fractures. One group of patients will undergo corrective surgery of the distal radius, with preoperative computer-assisted planning and virtual osteotomy, and the other group will undergo corrective surgery, with conventional (non-computer-assisted) preoperative planning. The investigators hypothesize that computer-assisted surgical planning will result in a better functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Extraarticular distal radius malunion requiring surgery
* Adult patient (> 18 yo)
* Fluent in English

Exclusion Criteria:

* Pregnant patient
* Prisoner
* Abnormal contralateral forearm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jupiter Jesse, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Leong NL, Buijze GA, Fu EC, Stockmans F, Jupiter JB; Distal Radius Malunion (DiRaM) collaborative group. Computer-assisted versus non-computer-assisted preoperative planning of corrective osteotomy for extra-articular distal radius malunions: a randomized controlled trial. BMC Musculoskelet Disord. 2010 Dec 14;11:282. doi: 10.1186/1471-2474-11-282. PMID 21156074

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Computer-Assisted Surgical Planning
Started | 20 | 20
Completed | 17 | 20
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Adult patients electing for corrective osteotomy for symptomatic extra-articular distal radial malunion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Computer-Assisted Surgical Planning | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (15.3) | 50.3 (19.6) | 51.2 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 1 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Disability of the Shoulder and Hand Score
Description: DASH score is a measure of upper extremity function. It ranges 0-100, where higher scores indication more disability and worse upper extremity function.
Time Frame: 0, 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | Computer-Assisted Surgical Planning
Number analyzed (Participants) | 17 | 20
Units on a scale
  0 months | 46.2 (25.0) | 51.8 (20.6)
  3 months | 27.9 (19.0) | 33.8 (24.0)
  6 months | 23.8 (18.9) | 24.1 (20.1)
  12 months | 22.8 (20.4) | 18.8 (18.0)

2. Secondary Outcome: Patient-Rated Wrist Evaluation (PWRE_
Description: PRWE score is a measure of wrist function. It ranges 0-100, where higher scores indication more disability and worse wrist function.
Time Frame: 0, 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | Computer-Assisted Surgical Planning
Number analyzed (Participants) | 17 | 20
Units on a scale
  0 months | 50.4 (20.1) | 58.2 (17.2)
  3 months | 28.7 (23.4) | 35.3 (28.7)
  6 months | 22.8 (16.7) | 22.8 (15.0)
  12 months | 22.3 (24.3) | 25.3 (20.6)

3. Secondary Outcome: Numerical Rating Scale for Pain
Description: Pain rated on a scale of 0-10, where 0 is no pain and 10 is severe pain
Time Frame: 0, 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | Computer-Assisted Surgical Planning
Number analyzed (Participants) | 17 | 20
Units on a scale
  0 months | 5.9 (2.8) | 6.2 (2.5)
  3 months | 2.4 (2.2) | 3.4 (2.3)
  6 months | 2.6 (2.8) | 3.2 (2.4)
  12 months | 2.1 (2.8) | 2.8 (2.1)

4. Secondary Outcome: Numerical Rating Scale for Satisfaction
Description: Satisfaction rated on a scale of 0-10, where 0 is not satisfied and 10 is completely satisfied
Time Frame: 0, 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | Computer-Assisted Surgical Planning
Number analyzed (Participants) | 17 | 20
Units on a scale
  0 months | 3.0 (1.7) | 2.8 (5.4)
  3 months | 8.4 (1.4) | 7.5 (2.0)
  6 months | 7.7 (2.2) | 7.6 (1.8)
  12 months | 8.4 (1.7) | 8.0 (1.9)

ADVERSE EVENTS:
Arm/Group | Control | Computer-Assisted Surgical Planning
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No